CLINICAL TRIAL: NCT05226286
Title: Evaluation of Implantable Tibial Neuromodulation Pivotal Study
Brief Title: Evaluation of Implantable Tibial Neuromodulation Pivotal Study (TITAN 2)
Acronym: TITAN 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20061
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Neoplasm Staging; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Medtronic Implantable Tibial Neuromodulation (TNM) System — Stimulation of the tibial nerve using Medtronic's tibial neuromodulation device.

SUMMARY:
The purpose of this prospective, multicenter study is to assess the safety and efficacy of tibial neuromodulation using the Medtronic Tibial Neuromodulation (TNM) system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older
2. Qualifying voiding diary
3. Have a diagnosis of UUI for at least 6 months
4. Failed and/or are not a candidate for conservative therapies.
5. Willing and able to accurately complete study diaries, questionnaires, attend visits, operate the system, and comply with the study protocol
6. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have primary stress incontinence
2. History of a prior implantable tibial neuromodulation system
3. Anatomical defects, clinically significant edema or previous surgeries which precludes use of the device
4. Previous pelvic floor surgery in the last 6 months
5. Women who are pregnant or planning to become pregnant during the course of the study
6. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
7. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mylene Champs, Study Director — Medtronic
Locations (29):
- United States (29):
  - Urology Centers of Alabama, Homewood, Alabama
  - Georgia Urology, Cartersville, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Providea Health Partners, Evergreen Park, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Chesapeake Urology Associates, Towson, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Minnesota Urology, Plymouth, Minnesota
  - Mayo Clinic Urology, Rochester, Minnesota
  - Summit Health Englewood, Englewood, New Jersey
  - Summit Health Voorhees, Voorhees Township, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Associated Medical Professionals, Syracuse, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Alliance Urology Specialists, Greensboro, North Carolina
  - FirstHealth Urogynecology, Hamlet, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Urology Surgeons of Oklahoma, Oklahoma City, Oklahoma
  - Prisma Health, Greenville, South Carolina
  - Sanford Female Pelvic Medicine & Reconstructive Surgery Clinic, Sioux Falls, South Dakota
  - Urology Partners of North Texas Research Institute, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Ascension Columbia St. Mary's, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects who signed the study-specific informed consent form (ICF) were considered enrolled in the study.
Groups:
- Enrolled Subjects: Eligible subjects who signed the study-specific informed consent form (ICF) were considered enrolled in the study.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started | 188
Implanted | 126
Day 7 | 126
Month 1 | 125
Month 2 | 125
Month 3 | 125
Month 6 | 125
Month 12 | 120
Month 24 | 104
Completed | 104
Not Completed | 84
Not completed — Screen failures prior to implant | 62
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Device explant with no planned replacement | 1
Not completed — Planned surgery with an implanted metal material closer than allowed in research protocol | 1
Not completed — Transitioned to urethral catheter/suprapubic tube | 1

BASELINE CHARACTERISTICS:
Population: All Implanted analysis set: Includes subjects who were implanted.
Groups:
- Implanted Subjects: Includes subjects who were implanted
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 108
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 126
BMI [Mean (Standard Deviation); unit: kg/m2] | 34.8 (8.61)

OUTCOME MEASURES:

1. Primary Outcome: UUI Responder
Description: Proportion of TNM subjects experiencing a reduction of 50% or more in daily urinary urge incontinence (UUI) episodes (UUI responder rate) at 6 months after device implant.
Time Frame: 6 months
Population: Includes subjects who were implanted and had data available at baseline and 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Implanted Subjects: Includes subjects who were implanted and had 6 month data available
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 123
Participants | 72

2. Secondary Outcome: UUI Change From Baseline
Description: Change in UUI episodes at 6 months compared to baseline in subjects with UUI at baseline.
Time Frame: 6 months
Population: Includes subjects who were implanted and had data available at baseline and 6 months
Measure: Mean (Standard Deviation); unit: UUI episodes (per day)
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 123
UUI episodes (per day) | -2.8 (3.12)

3. Secondary Outcome: UF Change From Baseline
Description: Change in daily UF episodes at 6 months compared to baseline in subjects with UF at baseline.
Time Frame: 6 months
Population: Includes subjects who were implanted and had data available at baseline and 6 months
Measure: Mean (Standard Deviation); unit: UF episodes (per day)
Groups:
- Subjects With Baseline UF: Urinary frequency (UF) subjects are those who have ≥ 10 urinary frequency episodes per day at baseline.
Arm/Group | Subjects With Baseline UF
Number analyzed (Participants) | 59
UF episodes (per day) | -2.6 (2.94)

4. Secondary Outcome: UPS Change at 6 Months
Description: Change in urinary urgency assessed through the UPS at 6 months compared to baseline.
  The UPS (Urgency Perception Scale) was developed to assess urgency associated with overactive bladder (OAB). The UPS is a single question assessed at each visit and has 3 options for responses: 1, 'I am usually not able to hold urine'; 2, 'I am usually able to hold urine until I reach the toilet if I go immediately'; and 3, 'I am usually able to finish what I am doing before going to the toilet'. Change from baseline is calculated by subtracting the baseline value from the follow-up value. Therefore, the change can range from -2 to 2 (with positive change indicating an improvement).
Time Frame: 6 months
Population: Includes subjects who were implanted and had data available at baseline and 6 months
Measure: Mean (Standard Deviation); unit: Score on Urgency Perception Scale
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 125
Score on Urgency Perception Scale | 0.4 (0.74)

5. Secondary Outcome: OAB-q Change From Baseline
Description: Change in Overactive Bladder Quality of Life Questionnaire (OAB-q) health related quality of life (HRQL) Total Score at 6 months compared to baseline.
  Details related to OAB-Q HRQL:
  OAB-q HRQL minimum value total score: 33 OAB-q HRQL maximum value total score:198 A positive change in OAB-q HRQL score represents an improvement.
Time Frame: 6 months
Population: Includes subjects who were implanted and had data available at baseline and 6 months
Measure: Mean (Standard Deviation); unit: OAB-q HRQL Total Score
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 125
OAB-q HRQL Total Score | 27.1 (25.79)

ADVERSE EVENTS:
Time Frame: AEs were collected throughout the study once the informed consent form was signed. This results section is showing the AEs that happened at or after implant through 24-month follow-up visit.
Description: For this study, all adverse events (AE) were collected regardless of relationship to the neurostimulator, external device, procedure, study aid, or therapy.
  Notes: The 1 death that happened in the Study was not related to the neurostimulator, external device, procedure, study aid, or therapy. Only 1 of the serious Adverse event was related (Clostridium difficile colitis).
Groups:
- Implanted Subjects: All Implanted analysis set: Includes subjects who were implanted
Arm/Group | Implanted Subjects
All-Cause Mortality (participants affected / at risk) | 1/126
Serious Adverse Events (participants affected / at risk) | 35/126
Other Adverse Events (participants affected / at risk) | 81/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Subjects (N=126)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Post procedural infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Marginal zone lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular node dysfunction (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Intestinal resection (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Subjects (N=126)
COVID-19 (Infections and infestations) | 30 (30)
Conjunctivitis (Infections and infestations) | 8 (8)
Nasopharyngitis (Infections and infestations) | 9 (10)
Urinary tract infection (Infections and infestations) | 36 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12)
Fall (Injury, poisoning and procedural complications) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT05226286/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT05226286/SAP_001.pdf